CLINICAL TRIAL: NCT03727243
Title: Molecular Diagnosis and Risk Stratification of Sepsis in India
Acronym: MARS-India
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Kasturba Medical College (Other); BioMérieux (Industry)
Responsible Party: Principal Investigator, W. J. Wiersinga, MD, Professor of Medicine, Chair division of Infectious Diseases and head of infectious diseases research group at the centre for experimental and molecular medicine (CEMM), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 371/2018
Record Dates: First submitted 2018-10-26; First posted 2018-11-01 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Sepsis; Septic Shock; Sepsis Syndrome
Keywords: Pneumonia; Infection; Tropical Infection; Endotypes; Biomarkers; Immunephenotyping; Lower middle-income countries (LMIC); Microbiome; Post-sepsis survival; Multi-omics
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome; Pneumonia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, RNA, DNA, PBMCs, Faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Septic/septic shock patients: Patients with underlying confirmed or probable cause of infection leading to sepsis or septic shock will form the active group of interest.
- Non-septic/sterile inflammation patients: Patient with severe trauma, severe burns and patients admitted to ICU after major surgery or pancreatitis. Active comparator group.
- Healthy control patients: Active comparator group.

SUMMARY:
Background: Globally, sepsis is common with an estimated population incidence of 437 cases per 100, 000 person-years and acute mortality of 26%, one of the few major medical conditions whose incidence and resulting mortality continues to rise. However, true burden is likely significantly higher as a recent meta- analysis could find no data from LMIC where 87% of the world's population resides.

Objective: Generate new knowledge that will eventually provide rapid and accurate information about an individual patient suffering from sepsis (or critical illness), including which type of microorganism is responsible for the infection and the severity and stage of the patient's immune response.

Methods: MARS-India will be a prospective longitudinal, single-centre observational study, conducted in mixed ICU's of a >2000 bedded tertiary teaching hospital in Manipal, India. The investigators will recruit to three groups- sex and age-matched healthy volunteers (n=150) and patients diagnosed with sepsis/septic shock or non-infectious ICU admissions such as severe trauma, severe burns and patients admitted to ICU after major surgery (n=400). The investigators have optimised a workflow to follow and describe the immunoinflammatory status of septic patients (as well as severe trauma/burn and major surgery) during the first 6 months after their initial injury. At fixed time points the investigators will collect blood in PaxGene, heparin, citrate and EDTA tubes in addition to routine bloods and microbiological samples. Rectal swabs and stool will also be taken for microbiome analysis. Immune functional tests will be performed to determine whole-blood cytokine/chemokine production in response to ex-vivo stimulation using an 8-panel assay. Additionally, complete immunophenotyping using flow cytometry including HLA-DR expression and lymphocyte subsets will be obtained.

DETAILED DESCRIPTION:
New sepsis 3.0 definition has for the first time included a dysregulated host response to infection as the cause of organ dysfunction, however, sepsis remains a highly heterogeneous syndrome without an accepted definition of what constitutes a dysregulated host response. The field is only now realising that inclusion of specific characteristics of the host response (transcriptomic or immunological profiles) facilitate stratification of patients with sepsis into subgroups (endotypes), allowing for prognostic enrichment and targeted therapeutic intervention.

Unfortunately, new guidelines continue to ignore the role of pathogens, virulence, sites of infection and lower-socio-economic settings. Additionally, it remains to be seen whether parasitic, viral and fungal conditions, common in LMIC, should be lumped with bacterial infections in the definition of sepsis. MARS -India will allow the investigators to compare these parameters and those of multi-drug resistant (MDR) pathogens on the impact of the host response and outcomes in sepsis. Not least develop an accurate temporal association of endotypes and detailed understanding of the immune suppressed phenotype. A functional immunology approach throughout and correlations with changes in the gut microbiome will further fortify our understanding of sepsis pathophysiology to help establish a 'sepsis fingerprint' and framework for novel interventions in future. Epidemiology data in itself will considerably heighten our understanding towards a global perspective on sepsis.

Furthermore, little guidance is offered in the Surviving Sepsis Guidelines toward optimal management of the seemingly cured post-acute sepsis patient, who is commonly readmitted with an infection or worse has a significantly reduced life expectancy (>40% 1yr mortality in some studies). MARS-India will also aim to establish the burden of this stage of sepsis in a LMIC setting and study the underpinning pathophysiology in more detail to establish groundwork in uncovering pathways for future therapeutic targeting.

It is apparent that biomarkers reflecting activity of targetable immunological pathways will be of paramount importance in managing the septic patient in future.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and over in the intensive care units of Kasturba Hospital, Manipal (and meeting the study population definitions below)
* Sepsis - defined as the presence of infection diagnosed within 24 hours of ICU admission with probable or definite likelihood, accompanied by organ dysfunction represented by an increase in the Sequential Organ Failure Assessment (SOFA) score of 2 points or more. Septic shock is defined as per the recent Sepsis 3.0 consensus guidelines.
* Serious trauma within 24 hours, with patient directly admitted to ICU (injury severity score (ISS) >15).
* Severe burns (total surface area burned >30%).
* Major surgery or pancreatitis/non-infectious inflammation.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients with a 'withdrawal of care' decision at time of inclusion
* Patients whose anticipated duration of hospitalisation in ICU is estimated <48 hours
* Extra-corporeal circulation in the month preceding inclusion in the case of cardiac surgery
* Patient with restricted liberty or under legal protection
* Expected lifespan <3 months due to pre-existing comorbidities
* Blood transfusion >4 units in past week
* Second admission to ICU or previous enrolment in study (within same hospital admission)
* Transfer from other hospital ICU (if greater than 24hrs in total)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in the general, emergency and neuro ICU's of Kasturba Hospital, Manipal. KMC hospital is a >2000 bedded tertiary care hospital that treats patients from a wide geographic area which can sometimes stretch beyond the state of Karnataka itself. Most patients will be from a mixture of urban and rural settings, with tropical infectious presentations varying throughout the year.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-06-11 (Estimated)

PRIMARY OUTCOMES:
Molecular information of individual host-pathogen response and outcomes in sepsis. | 2 years
  Using RNA sequencing the investigators will map the transcriptional picture of sepsis in a tropical LMIC setting and also map the changes longitudinally.
Gut microbiome alterations in correlation to sepsis endotypes and associated post sepsis mortality/re-admission. | 3 years
  This will make use of 16S PCR and shotgun metagenomic sequencing.

SECONDARY OUTCOMES:
Quantify mortality, morbidity and re-admissions in sepsis survivors from a LMIC setting. | 2.5 years
  Patients surviving sepsis will be followed up for 6 months post discharge.
Stratification of septic patients by severity and type of immune response to infection. | 3 years
  This will utilise a multi-omics approach and up-to-date bioinformatic techniques to bring together the previous outcomes with functional immunology profiles. Ultimate aim will be to generate a novel biomarker panel.

CONTACTS AND LOCATIONS:
Overall Officials: Chiranjay Mukhopadhyay, MD, Phd, Principal Investigator — Associate Dean and Professor Department of Microbiology, KMC Manipal; Willem Joost Wiersinga, MD, PhD, Principal Investigator — Professor of Medicine, Chair Devision of Infectious Diseases and head of infectious diseases research group at the centre for experimental and molecular medicine (CEMM), Amsterdam UMC (AMC); Tom van der Poll, Principal Investigator — Professor of Medicine and Chair department of Medicine, Amsterdam UMC (AMC)
Locations (1):
- Kasturba Hospital, Kasturba Medical College (KMC), Manipal Academy of Higher Education (MAHE), Udupi, Karnataka, India

REFERENCES:
- [Derived] Virk HS, Biemond JJ, Earny VA, Chowdhury S, Frolke RI, Khanna SM, Shanbhag V, Rao S, Acharya RV, Balakrishnan JM, Eshwara VK, Varma MD, van der Poll T, Wiersinga WJ, Mukhopadhyay C. Unraveling Sepsis Epidemiology in a Low- and Middle-Income Intensive Care Setting Reveals the Alarming Burden of Tropical Infections and Antimicrobial Resistance: A Prospective Observational Study (MARS-India). Clin Infect Dis. 2025 Feb 5;80(1):101-107. doi: 10.1093/cid/ciae486. PMID 39352692